CLINICAL TRIAL: NCT02250027
Title: A Multicenter, Randomized, Double-blind, Parallel Group Study to Determine the Optimal Dose of HL301 After 7 Days Oral Administration in Acute Bronchitis or Acute Exacerbations of Chronic Bronchitis Patients (HL301: Mixed Extract of Rehmannia Glutinosa, Schisandra and so on)
Acronym: HL301
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_HL301_201
Record Dates: First submitted 2014-09-02; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Acute Bronchitis; Acute Exacerbations of Chronic Bronchitis
Keywords: acute bronchitis; acute exacerbations of chronic bronchitis
MeSH Terms: conditions — Bronchitis | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- experimental A (0.6g/day) (Experimental): HL301 0.6g/day: 2 capsules at once, 3 times a day, for 7 days
  Interventions: Drug: HL301 300mg capsule; Drug: Placebo
- experimental B (1.2g/day) (Experimental): HL301 1.2g/day: 2 capsules at once, 3 times a day, for 7 days
  Interventions: Drug: HL301 300mg capsule; Drug: Placebo
- experimental C (1.8g/day) (Experimental): HL301 1.8g/day: 2 capsules at once, 3 times a day, for 7 days
  Interventions: Drug: HL301 300mg capsule
- Placebo (Placebo Comparator): placebo: 2 capsules at once, 3 times a day, for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HL301 300mg capsule — 2 capsules at once, 3 times a day, for 7 days
  Other Names: experimental A (0.6g/day) : HL301 300mg 2 capsule; experimental B (1.2g/day) : HL301 300mg 4 capsule; experimental C (1.8g/day) : HL301 300mg 6 capsule
  Arms: experimental A (0.6g/day); experimental B (1.2g/day); experimental C (1.8g/day)
Drug: Placebo — 2 capsules at once, 3 times a day, for 7 days
  Other Names: Microcrystalline Cellulose
  Arms: Placebo; experimental A (0.6g/day); experimental B (1.2g/day)

SUMMARY:
The purpose of this study is to determine the optimal dose of HL301 in patients with acute bronchitis or acute exacerbations of chronic bronchitis.

- BSS(Bronchitis Severity Score), BCSS(Breathlessness, Cough, and Sputum Scale), evaluation of symptoms of cough and sputum

ELIGIBILITY:
Inclusion Criteria:

1. Both gender, 19 years ≤ age ≤ 80 years
2. Acute bronchitis or acute exacerbations of chronic bronchitis patients with BSS(Bronchitis Severity Score)* ≥ 5point at Visit1 and Visit2
3. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Patients who were increased the bleeding tendency
2. Patients with any of Alanine aminotransferase, Aspartate aminotransferase or serum Blood Urea Nitrogen, Creatinine> 2 times of the normal upper range
3. Patients who investigators determines to severe respiratory disease that would interfere with study assessment
4. Patients with COPD(Chronic Obstructive Pulmonary Disease) history of stage 3 or more
5. Patients who were treated with oral systemic adrenocortical hormone or immunosuppressive drug within 4 weeks prior to study participation
6. Patients who were treated with oral β2-agonist, anticholinergic, Methylxanthine, antibiotics, antihistamines, sympathomimetic agent or oriental medicine/health functional food for antitussive and mucolytic Effect within 1 weeks prior to study participation
7. Patients who were treated with oral Antitussive, Mucolytic Agents,systemic antimicrobial agent within 3 days prior to study medication dosing
8. Patients with drug or alcohol abuse
9. Patients with clinically significant active liver, renal, cardiovascular, respiratory, endocrine, central nervous system disease or history of malignant tumor or mental illness(except no relapse for 5 years after surgery)
10. The aged person with severe medical history which is mental disorder(dementia), cancer, chronic renal failure, chronic liver failure
11. Pregnant or breast-feeding
12. Patients currently participating in or has participated in other clinical study within 30 days prior to study participation
13. Patients who investigators determines not appropriate to take part in this clinical study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Bronchitis Severity Score | baseline(day 0) and day 7
  Bronchitis Severity Score

SECONDARY OUTCOMES:
Breathlessness, Cough, and Sputum Scale | baseline(day 0) and day 7
  Breathlessness, Cough, and Sputum Scale
evaluation of symptoms of cough and sputum | baseline(day 0) and day 7
Total usage of acetaminophen | baseline(day 0) and day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea